CLINICAL TRIAL: NCT07334548
Title: A Comparative Analysis of Polypropylene Conventional Mesh Fixation Versus 3-point Fixation Technique to Assess Post-Surgical Outcomes in Lichtenstein Hernia Repair (RCT).
Brief Title: Post-Surgical Outcomes of Conventional vs 3-Point Mesh Fixation in Lichtenstein Repair: An RCT
Acronym: COMET
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Bushra shirazi, Professor, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIUT-ERC-2025/A-573
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: İnguinal Hernia; Complication,Postoperative; Pain, Postoperative
Keywords: comparision; lichtenstein mesh repair; 3-point fixation; inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal; Postoperative Complications; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Mesh Fixation Group (Standard Fixation (Active Comparator): Lichtenstein inguinal hernia repair with polypropylene mesh fixed using the conventional technique (multiple non-absorbable sutures across the inguinal floor) to measure Immediate postoperative complications: seroma, hematoma, wound infection, acute pain (post-op days 1 and 7) and long-term outcomes: chronic groin pain (CGP) and hernia recurrence (3 months and 6 months follow-up)
  Interventions: Procedure: Conventional Mesh Fixation
- 3-Point Mesh Fixation Group (Minimal Fixation) (Experimental): Lichtenstein inguinal hernia repair with polypropylene mesh fixed at only three strategic points to minimize tissue trauma. To measure Immediate postoperative complications: seroma, hematoma, wound infection, acute pain (post-op days 1 and 7) and long-term outcomes: chronic groin pain (CGP) and hernia recurrence (3 months and 6 months follow-up)
  Interventions: Procedure: 3-point mesh fixation

INTERVENTIONS:
Procedure: 3-point mesh fixation — Patients in this group will undergo Lichtenstein hernia repair with polypropylene mesh fixed at three key points only (pubic tubercle, inguinal ligament and conjoint tendon). The fixation points will be strategically chosen to provide sufficient stability while minimizing tissue trauma.
  Rationale: Reducing the number of fixation points is expected to decrease the risk of nerve entrapment, muscle irritation, and post-operative pain, without compromising mesh position or increasing recurrence rates
  Arms: 3-Point Mesh Fixation Group (Minimal Fixation)
Procedure: Conventional Mesh Fixation — Patients in this group will undergo Lichtenstein tension-free hernia repair using a polypropylene mesh secured with the conventional technique. Multiple non-absorbable sutures will be placed across the inguinal floor to anchor the mesh between the transversalis fascia and the external oblique aponeurosis
  Arms: Conventional Mesh Fixation Group (Standard Fixation

SUMMARY:
This is a single-center, parallel-group randomized controlled trial conducted in 2025-2025 at the General Surgery Ward of the Sindh Institute of Urology and Transplantation (SIUT), Karachi. This study shows the comparative analysis of polypropylene conventional mesh fixation versus 3-point fixation technique to assess Post-Surgical Outcomes in Lichtenstein Hernia Repair

DETAILED DESCRIPTION:
This randomized controlled trial is designed to compare the outcomes of conventional mesh fixation versus 3-point fixation in patients undergoing Lichtenstein inguinal hernia repair. The primary focus is to evaluate immediate postoperative outcomes-pain, seroma, hematoma, and wound infection-on postoperative days 1 and 7. Long-term outcomes, including recurrence and chronic groin pain, will be assessed at 3 months and 6 months. The study will include 64 patients aged 18-70 years, meeting ASA I-II criteria, and presenting with unilateral inguinal hernia. They will be randomly assigned to one of the two fixation techniques under a single-blind design where only the patient is blinded.

Data will be collected using a structured proforma capturing demographics, perioperative findings, and postoperative follow-up information. Pain will be measured using the Visual Analog Scale (VAS) with standardized analgesia. Data analysis will be performed using SPSS, with appropriate statistical tests applied according to the nature of the variables. A significance level of p < 0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to the outpatient department with unilateral inguinal hernia requiring Lichtenstein repair

Age between 18-70 years Both male and female ASA I-II

Exclusion Criteria:

Recurrent, bilateral, complicated, or incisional hernia Patients with pre-existing obstructive LUTS Chronic kidney disease (CKD), patients on hemodyalysis. Chronic liver disease (CLD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Acute post operative pain | 7 days
  Acute Postoperative pain measured using the Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst pain imaginable).
  Standard analgesia (ketorolac 30 mg twice daily) will be provided.
wound infection | 7- 14 days
  Defined according to CDC criteria: redness, warmth, discharge, or systemic signs of infection at the incision site
Seroma | 7-14 days
  The fluid collection at the surgical site which will be confirmed clinically or by ultrasound if needed.
hematoma | 7 days
  A localized collection of blood at the operative site which will be assessed clinically for swelling, discoloration, and need for intervention.

SECONDARY OUTCOMES:
Chronic groin pain | 6 months
  Pain persisting beyond three months post-surgery, measured using VAS and patient-reported impact on daily activities.
  Severity categorized as mild, moderate, or severe.
Hernia recurrence | 6 months
  Recurrence of previously repaired inguinal sweling/hernia clinically diagnosed by physical examination and confirmed with ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan